CLINICAL TRIAL: NCT05669742
Title: Evaluating the Safety and Efficacy of Empagliflozin Addition in Modulating Metabolic Disturbances Associated With Olanzapine in Schizophrenia Patients.A Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: Empagliflozin Addition in Modulating Metabolic Disturbances Associated With Olanzapine in Schizophrenia Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Elberri, Lecturer of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMPA2022
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sodium-glucose Transport Protein Two Inhibitor (SGLT2),Metabolic Deficits Caused by Antipsychotics
MeSH Terms: interventions — empagliflozin; Olanzapine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 as control group (Active Comparator)
  Interventions: Drug: olanzapine
- Group two as Empagliflozin (Active Comparator)
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — sodium-glucose transport protein two inhibitor
  Arms: Group two as Empagliflozin
Drug: olanzapine — antipsychotics
  Arms: Group 1 as control group

SUMMARY:
Olanzapine is a thieno-benzodiazepine derivate that is effective managing the symptoms of schizophrenia and reducing the psychopathological symptoms of psychosis. It is also effective in controlling the acute manic episodes associated with bipolar disorder, and have provided some therapeutic advantages over other antipsychotic agents (Citrome et al., 2019).

However, Ola administration has been reported to induce profound BWG accompanied with higher incidence of metabolic deficits, such as hypertension, diabetes and hyperlipidemia, as compared to other antipsychotic agents (Mauri et al., 2014).

Adjunctive treatment with other agents that can minimize or normalize Ola-induced BWG can enhance the safety and tolerability profiles of an effective antipsychotic, thus highlighting the need to develop improved therapies or interventions to minimize these side effects. A meta-analysis of 12 published studies found that antidiabetic drugs such as metformin improved metabolic parameters in patients treated with antipsychotics (de Silva et al., 2016).

These studies encouraged the evaluation of other antidiabetic agents as adjunctive therapies to minimize Ola-induced BWG. Empagliflozin (EMPA)is the third-generation anti-diabetic drug acting as sodium-glucose transport protein two inhibitor (SGLT2), which provides a new mechanism of action to improve glycemic control with modest decreases in systolic blood pressure and body weight (Pradhan et al., 2019). The effects of EMPA on Ola-induced BWG have not been determined and require further investigation.

ELIGIBILITY:
Inclusion Criteria:

Schizophrenia Patients treated with Olanzapine with ages ranging from 18 to 60 years.

Exclusion Criteria:

patients who had any other inflammatory disease (cardiovascular, asthma, bone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight and body mass index (BMI) | up to 12 weeks
  a person's weight in kilograms (or pounds) divided by the square of height in meters and measure of body fat based on height and weight that applies to adult men and women body mass index = wt (kilogram) divideed by height in meter square

SECONDARY OUTCOMES:
Adverse events (AE) as measures of safety and tolerability of Empagliflozin | up to 12 weeks
  any side effects of the used intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt